CLINICAL TRIAL: NCT02904811
Title: Prevention of Diseases Induced by Chlamydia Trachomatis
Acronym: i-PREDICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Reference Center (NRC) for Chlamydia infections, UMR1181 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P150950; AOM 15-0063 (Other: AP-HP)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Genital Chlamydia Trachomatis Infection
Keywords: Chlamydia trachomatis; Pelvic inflammatory disease
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Testing for Ct infection immediately
  Participants will perform self-taken vaginal samples.
  The positive results for Ct will be examined and treated and their partner will also be informed to do so.
  Interventions: Other: Testing for Ct infection immediately
- Control group (Experimental): Testing for Ct infection at the end of the study
  Interventions: Other: Testing for Ct infection at the end of the study

INTERVENTIONS:
Other: Testing for Ct infection immediately — Self-taken vaginal samples will be immediately tested for Ct infection at the National Reference Centre (CNR) at University of Bordeaux, using a commercially available CE marketed real-time PCR assay.
  Arms: Intervention group
Other: Testing for Ct infection at the end of the study — Self-taken vaginal samples will be tested for Ct infection at the end of the study (M18).
  Arms: Control group

SUMMARY:
The main objective of the study is to determine whether early screening and treating young women (<25 years of age) for genital Chlamydia Trachomatis (Ct) infection reduces the cumulative incidence of pelvic inflammatory disease (PID) over 24 months.

As secondary objectives, the study aims

* To determine the baseline prevalence and the incidence of Ct infection;
* To improve knowledge on natural history of Ct infection in young women such as the rate and timing of progression to PID (at the beginning of the infection, at the end, throughout the course of infection), as well as the incidence of reinfections with Ct;
* To investigate the relation between host immuno-genetic factors and the clearance, persistence and development of late complications (PID) as an explanation for the inter-individual heterogeneity in the susceptibility to and course of Ct infection.

DETAILED DESCRIPTION:
In this research project, the study aims to assess a screening strategy (early screening and treatment of Ct genital infection in young women to prevent complications) that may be implemented in the future if proved efficient 7 centers are involved in the enrollment (university health services), and 4 centers will participate in the study within the frame of the follow-up and final visit (hospital gynaecology departments).

Participants included will have to perform 4 self-taken vaginal samples linked to four online corresponding questionnaires, at different timeframes 6-month apart to each other (M0, M6, M12, M18). The first sampling (M0) will be performed at the university health service, this self-taken sampling could also be performed at home later in case of menstruation; the others (M6, M12, M18) will be performed at home (or at the university if problem of sampling kits receiving at home).

Participants will be randomly assigned to one of the two following arms:

* in the non-intervention arm, participants will follow current guidelines of Ct screening (i.e. opportunistic screening only in STI clinics for women aged less than 25 years old), and their samples will be tested for Ct at M18 by the NRC;
* in the intervention arm, analyses for Ct will be carried out immediately by the NRC.

A final visit with a hospital gynecologist is planned for all participants between M18 and M24 and aims at providing an extensive clinical examination to seek for potential signs of pelvic inflammatory disease and to treat participants if needed.

Based on all data collected on the electronic platform through questionnaires from the different visits, independent experts blinded on chlamydia status will assess PID status of all participants (no PID, probable PID, confirmed PID).

The duration of enrollment is planned for 36 months.

The duration of follow-up for each patient is 18 months to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* female students visiting the preventive medical centers of universities or the Ct screening test centers who participate in the study;
* participate in or will participate in the "i-Share" cohort;
* aged between 18 to 24 years,
* had prior sexual relations,
* written informed consent signed,
* affiliated to the social security bodies.

Exclusion Criteria:

* Known pregnancy.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1092 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence | At 24 months
  Cumulative incidence of first PID

SECONDARY OUTCOMES:
Incidence of first Ct infection | Up to 24 months
  Incidence of first Ct infection for negative participants at baseline
Duration of Ct infection | Up to 24 months
Proportion of Ct infection progressing to PID | Up to 24 months
Time of Ct infection progressing to PID | Up to 24 months
Proportion of spontaneous resolution of Ct infections | Up to 24 months
  Proportion of spontaneous resolution of Ct infections
Incidence of reinfections | Up to 24 months
  Incidence of reinfections

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Delarocque-Astagneau, MD, Study Chair — Université de Versailles Saint Quentin
Locations (1):
- Université de Versailles Saint Quentin, Versailles, Saint-Quentin-en-Yvelines, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tamarelle J, Thiebaut ACM, de Barbeyrac B, Bebear C, Bourret A, Fauconnier A, Ravel J, Delarocque-Astagneau E; i-Predict study group. Vaginal microbiota stability over 18 months in young student women in France. Eur J Clin Microbiol Infect Dis. 2024 Dec;43(12):2277-2292. doi: 10.1007/s10096-024-04943-3. Epub 2024 Sep 20. PMID 39302529
- [Derived] Tamarelle J, Thiebaut ACM, Sabin B, Bebear C, Judlin P, Fauconnier A, Rahib D, Meaude-Roufai L, Ravel J, Morre SA, de Barbeyrac B, Delarocque-Astagneau E; i-Predict study group. Early screening for Chlamydia trachomatis in young women for primary prevention of pelvic inflammatory disease (i-Predict): study protocol for a randomised controlled trial. Trials. 2017 Nov 13;18(1):534. doi: 10.1186/s13063-017-2211-1. PMID 29132441